CLINICAL TRIAL: NCT02783105
Title: Effects of Early Musical Intervention on Prevalence and Severity of Paroxysmal Sympathetic Hyperactivity After Severe Traumatic Brain Injury: the Prospective Randomized MUSIC-TCNV Trial.
Brief Title: Effects of Early Musical Intervention on Prevalence and Severity of Paroxysmal Sympathetic Hyperactivity After Severe Traumatic Brain Injury
Acronym: MUSIC-TCNV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion difficulties
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Fondation Apicil (Other); MDMS (Unknown); Association française des traumatisés crâniens d'Alsace (Unknown); Association strasbourgeoise des médecins et infirmiers en anesthésie réanimation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 6224
Record Dates: First submitted 2016-05-23; First posted 2016-05-26 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2016-11

CONDITIONS: Paroxysmal Sympathetic Hyperactivity
Keywords: Music therapy; Paroxysmal sympathetic hyperactivity; Traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Musical intervention (Experimental): Music is provided through headphones: Two 30-min musical sessions per day (one in the morning and one in the evening) beginning at the onset of desedation (Day 0) until day 21.
  Both have inverted "U" shape.
  Interventions: Other: Musical intervention
- Control (Sham Comparator): Patients wear headphones twice a day during 30 minutes, starting at the onset of desedation (Day 0) until day 21, but no music is provided (blank playlist): Sham
  Interventions: Other: Control

INTERVENTIONS:
Other: Musical intervention
  Arms: Musical intervention
Other: Control — Patients wear headphones twice a day during 30 minutes, starting at the onset of desedation (Day 0) until day 21, but no music is provided (blank playlist): Sham
  Arms: Control

SUMMARY:
Paroxysmal sympathetic hyperactivity (PSH) is a frequent symptom after traumatic brain injury and concerns up to 30% of severely brain-injured patients.

PSH is due to unbalanced autonomic nervous system activity, resulting in sympathetic surges causing hypertension, tachycardia, sweating and hypertonia. The affected patients suffer more pain, more cardiovascular distress, more infections and prolonged rehabilitation and mechanical ventilation; additionally it could lead to a worse outcome.

Classical music was shown to reduce autonomic nervous system imbalance in healthy people and in many medical diseases. It could be a means to dampen sympathetic surges for brain-injured patients presenting with PSH, as well.

Our study aims at demonstrating that early musical intervention, started with the weaning of sedation, can reduce both the prevalence and the severity of paroxysmal sympathetic hyperactivity in traumatic brain-injured patients.

ELIGIBILITY:
Inclusion Criteria:

* Severe traumatic brain injury (either initial Glasgow Coma Scale < 8 or intracranial pressure > 20mmHg for more than 20 min)
* National health service coverage
* Informed consent signed by next of kin

Exclusion Criteria:

* Non-traumatic brain injury
* Conditions interfering with measures: bilateral fixed pupils, temporal bone fracture including acoustic channel, eye trauma, previous eye surgery, otorrhagia, hypoacusis,
* Preexisting autonomic nervous system imbalance: severe diabetes, arrhythmias, pace maker, implantable defibrillator, cardiac transplantation
* Respiratory rate < 9/min
* Patient subject to guardianship or wardship
* Pregnant or breastfeeding woman
* Current participation in another biomedical research protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-11-20 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Paroxysmal Sympathetic Hyperactivity Assessment Measure [PSH-AM] (ranging from 0 to 29) | from desedation (Day 0) to Day 21.
  The PSH-AM combines the sum of Clinical Features Scale [CFS] (from 0 to 18) and the Diagnostic Likelihood tool [DLT] (from 0 to 11)

SECONDARY OUTCOMES:
Area under the Clinical Features Scale curve | from Day 0 to Day 21.
Mean Analgesia Nociception Index | from Day 0 to Day 21.
Neurological Pupil Index | from Day 0 to Day 21.
Pain (Critical-Care Pain Observation Tool) | from Day 0 to Day 21.
Neurological outcome (Wessex Head Injury Matrix) | from Day 0 to Day 21.
PSH-AM | Six and twelve months
Disability Rating Scale | Six and twelve months

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie Réanimation- Hôpital de Hautepierre, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No